CLINICAL TRIAL: NCT05441709
Title: Clinically Integrated Breastfeeding Peer Counseling to Promote Breastfeeding Equity
Brief Title: Furthering Equity Through Infant Feeding EDucation and Support
Acronym: FEEDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Northwestern University (Other); University of Chicago (Other); Rush University (Other)
Responsible Party: Principal Investigator, Ann Borders, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH20-406
Record Dates: First submitted 2022-06-15; First posted 2022-07-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Peer Counseling; Lay health worker; Infant Feeding
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to either standard lactation care or to standard lactation care plus clinically-integrated breastfeeding peer counseling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard lactation care is provided by postpartum RNs on the inpatient unit and RNs who are board certified in lactation (IBCLCs).Postpartum RNs provide support to all patients post delivery with direct breastfeeding, breast pump use, and addressing routine breastfeeding concerns. IBCLCs provide direct lactation care for more complicated lactation problems and is delivered in a dosed manner based on the nature of the lactation problem, with low-risk patients often having no encounters.
- ci-BPC with Standard of Care (Active Comparator): In addtion to normal standard of care (as described above), patients will also receive clinically-integrated breastfeeding peer counseling (ci-BPC) from a Peer Counselor at four timepoints throughout the perinatal period. The encounters will take place either in person or virtually and include: an intake encounter between 2- and 30 weeks gestation, a dedicated prenatal infant feeding education encounter, at least one inpatient encounter post-delivery during the delivery admission, and at least one postpartum encounter. Patients will also have access to a "warmline" that will include phone follow up by the next business day.
  Interventions: Behavioral: Ci-BPC with Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Ci-BPC with Standard of Care (SOC) — Clinically-integrated breastfeeding peer counseling (ci-BPC) is a practice that, supports the patient and the clinical care team by delivering culturally-appropriate breastfeeding help to motivate breastfeeding initiation, intensity, and duration, inspiring confidence for patients to set breastfeeding goals and meet them. ci-BPC is delivered by community health workers who have breastfed an infant, and have received basic training in breastfeeding support through a qualified BPC training organization. For this project, the Peer Counselor will make initial contact to patients randomized into the treatment arm via phone to schedule the Intake Encounter between 20 and 30 weeks gestation. Subsequently, each patient will receive a minimum of 3 additional encounters which can occur virtually or in-person. Patients randomized to the ci-BPC arm are additionally offered access to a "warmline" where messages will be returned by the next business day.
  Arms: ci-BPC with Standard of Care

SUMMARY:
The purpose of this study is to identify whether adding clinically integrated breastfeeding peer counseling (ci-BPC) to standard lactation care is associated with a reduction in disparities in breastfeeding intensity and duration for Black and Hispanic/Latine families.

DETAILED DESCRIPTION:
FEEDS is a randomized control trial comparing standard lactation care to standard lactation care plus a ci-BPC. This trial will take place at three hospitals in the Chicago land area, Swedish Hospital, Highland Park Hospital, and University of Chicago Medicine Hospital. The aims of the study are: (1) To determine whether ci-BPC reduces disparities in breastfeeding outcomes for Black and Hispanic/Latine participants, (2)To determine whether ci-BPC improves breastfeeding knowledge, attitude, access to support, and empowerment, (3) To understand implementation outcomes, facilitators, and barriers, and (4) To identify associated patient centered costs.

ELIGIBILITY:
Inclusion Criteria:

* 12 and 24 weeks gestation
* English or Spanish speaking
* Planning to parent their infant
* Planning to deliver at SH, HPH or UCM
* No prior exposure to ci-BPC

Exclusion Criteria:

* considering pregnancy termination or adoption
* Prior exposure to ci-BPC

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 990 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding duration | 6 weeks postpartum
  Total length of time in weeks that breastmilk feeds were provided to the infant, collected via participant self-report.
Breastfeeding duration | 6 months postpartum
  Total length of time in weeks that breastmilk feeds were provided to the infant, collected via participant self-report.

SECONDARY OUTCOMES:
Breastfeeding intensity-inpatient | During Delivery Admission
  Proportion of infant feedings during the delivery admission that are breastmilk only. Number of breastmilk feeds will be divided by the total number of infant feedings.
Breastfeeding intensity-post discharge | 6 weeks postpartum
  Proportion of infant feedings that are breastmilk only. Intensity will be calculated as # breastmilk feeds/day divided by total number of infant feedings/day as recorded in the infant feeding logs completed by study participants.
Breastfeeding intensity-post discharge | 6 months postpartum
  Proportion of infant feedings that are breastmilk only. Intensity will be calculated as # breastmilk feeds/day divided by total number of infant feedings/day as recorded in the infant feeding logs completed by study participants.

OTHER OUTCOMES:
Breastfeeding knowledge | Baseline 12-20 weeks
  Breastfeeding Knowledge Questionnaire, and questions regarding behavioral norms around breastfeeding
Breastfeeding knowledge | 6 weeks postpartum
  Breastfeeding Knowledge Questionnaire, and questions regarding behavioral norms around breastfeeding
Breastfeeding knowledge | 6 months postpartum
  Breastfeeding Knowledge Questionnaire, and questions regarding behavioral norms around breastfeeding
Infant feeding attitude- Iowa Infant Feeding Attitude Scale (IIFAS) | Baseline 12-20 weeks
  The Iowa Infant Feeding Attitudes Scale; 26 items with a 5 point likert scale, half of which measure favorability towards breastfeeding and the remaining half measuring favorability towards formula feeding, higher scores reflect positive attitudes towards breastfeeding and lower scores reflect positive attitudes towards formula.
Ci-BPC related costs | 6 weeks postpartum
  The time spent in BPC inpatient encounters, outpatient/telehealth appointments and support group sessions, travel time for BPC appointments, transportation for BPC appointments, and cellular data for telehealth BPC appointments.
Out of pocket cost | 6 weeks postpartum
  Supplies purchased for infant feeding, including breastfeeding supplies (e.g., pump and parts, storage, contained, bras, breast pads, billows), bottles, formula, and addition food cost (including supplements)
Feeding related opportunity costs | 6 weeks postpartum
  Time spent feeding infants (preparation, feeding, and clean up) for type of feeding (breast milk at breast, breast milk by bottle, formula)
Infant feeding attitude- Iowa Infant Feeding Attitude Scale (IIFAS) | 6 weeks postpartum
  The Iowa Infant Feeding Attitudes Scale; 26 items with a 5 point likert scale, half of which measure favorability towards breastfeeding and the remaining half measuring favorability towards formula feeding, higher scores reflect positive attitudes towards breastfeeding and lower scores reflect positive attitudes towards formula.
Infant feeding attitude- Iowa Infant Feeding Attitude Scale (IIFAS) | 6 months postpartum
  The Iowa Infant Feeding Attitudes Scale; 26 items with a 5 point likert scale, half of which measure favorability towards breastfeeding and the remaining half measuring favorability towards formula feeding, higher scores reflect positive attitudes towards breastfeeding and lower scores reflect positive attitudes towards formula.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Borders, MD, MS, Principal Investigator — Endeavor Health (NorthShore University HealthSystem)
Locations (4):
- United States (4):
  - Swedish Hospital, Chicago, Illinois
  - UChicago Medicine Hospital (University of Chicago), Chicago, Illinois
  - Endeavor Health (NorthShore University HealthSystem), Evanston, Illinois
  - Highland Park Hospital, Highland Park, Illinois

REFERENCES:
- [Derived] Keenan-Devlin LS, Smart BP, Hirschhorn L, Meier P, Jefferson U, Solomonides A, Wang CE, Handler A, Silver RK, Borders AEB. Clinically Integrated Breastfeeding Peer Counseling to Promote Breastfeeding Equity. Am J Perinatol. 2024 May;41(S 01):e2313-e2325. doi: 10.1055/s-0043-1771255. Epub 2023 Jul 21. PMID 37494586